CLINICAL TRIAL: NCT02560896
Title: Genomic Incidental Findings Disclosure (GIFD) in a Cancer Biobank: An Ethical, Legal and Social Implications (ELSI) Experiment (Protocol for Aim 3 Intervention)
Brief Title: Understanding Genetic Incidental Findings in Your Family (UNIFY Study)
Acronym: UNIFY
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 15-001209
Record Dates: First submitted 2015-08-27; First posted 2015-09-25 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Familial Pancreatic Cancer
Keywords: Family; History; Pancreas; Cancer; Genetic
MeSH Terms: conditions — Pancreatic carcinoma, familial; Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Currently, there is no clear legal or ethical guidance about how researchers and IRBs ought to proceed when the research participant in a biobank is deceased and there is clinically relevant information that could be disclosed to family members. This study is designed to test a procedure offering genetic information to family members of research participants who participated in a pancreatic cancer biobank in a Health Insurance Portability and Accountability Act (HIPAA) -compliant design.

DETAILED DESCRIPTION:
To develop, prototype, and evaluate a novel procedure for offering probands' genetic results to family members. The intervention is to offer a deceased research participant's actionable germline genetic research finding, and depending upon the choice made by the next of kin, a disclosure of the research finding by a genetic counselor in a family conference call. Using mixed methods (quantitative and qualitative), the investigators will assess decision making, family communication, and actions and responses in individuals from families in which a proband is known to have a deleterious germline mutation in one of several known cancer susceptibility genes.

ELIGIBILITY:
Family members and others authorized to receive health information of participants enrolled under Institutional Review Board (IRB) #354-06 and #355-06 who carry one of several known cancer susceptibility genes.

* Mentally competent and able to provide informed consent
* Able to understand and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Familial Pancreatic Cancer Kindred
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Uptake of disclosure invitation | 6 months
  The primary outcome is: relative proportions of individuals who, when offered genetic results of a deceased family member who participated in a biobank study, will decide to learn those results. Uptake will be a binary outcome (Yes/No). We will enumerate the number of invited participants who choose to learn results and who choose not to learn results.

SECONDARY OUTCOMES:
Frequency and duration of physical activity | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: number of self-reported days per week and exercise duration(minutes).
Frequency and duration of alcohol use | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: number of drinks containing alcohol taken per week over previous six months; frequency drinking 6 or more drinks in one occasion in past 6 months (Never; Less than monthly; Monthly; 2 to 3 times per week; 4 or more times per week)
Current cigarette smoking status | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: Current cigarette smoker (Yes/No)
Quality and amount of sleep | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: Quality of sleep (Very good; Fairly good; Fairly bad; Very bad); Number of hours of sleep in a 24 hour period (hours and minutes)
Frequency of fruit and vegetable consumption | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: Number of servings eaten in a typical day (None; 1 or less; 2; 3; 4; 5 or more)
Frequency of red meat consumption | 6 months
  We will measure and compare changes between baseline and 6 months following genetic test disclosure: Number of times consumed per typical week (0; 1 to 5; 6 to 10; 11 to 15; 16 to 20; 21 or more).
Uptake of genetic testing | 6 months
  The relative proportion of individuals who request and obtain genetic testing on their own by 6 months
Quality of life | 6 months
  Changes in self-reported quality of life on a scale of 0(a bad as it can be) to 10 (as good as it can be)
Perceived cancer risk/worry | 6 months
  Changes in self-reported worry of developing cancer on a scale of 1 (not at all or rarely to 4 (almost all the time)
Decision regret | 6 months
  Self-reported rating of regret to learn/not learn their relative's genetic research result using a 5-item scale rating (Strongly agree to Strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Petersen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials